CLINICAL TRIAL: NCT06080737
Title: Effects of Awake Prone Positioning on Long-term Quality of Life in Patients Managed in the ICU Under Nasal High Flow for SARS-CoV2 Pneumonia, a Cohort Study Nested Within a Randomized Trial
Brief Title: Long Term Effects of Awake Prone Positioning in COVID-19 ICU Patients
Acronym: Long-termAPP
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: DR 230170 - Long-term APP
Record Dates: First submitted 2023-10-10; First posted 2023-10-12 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: SARS-CoV 2 Pneumonia
Keywords: long-term quality of life; awake prone positioning; acute respiratory distress syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- standard oxygen group: telephone interview comprising a quality of life questionnaire
  Interventions: Other: quality of life questionnaire
- awake prone group: telephone interview comprising a quality of life questionnaire
  Interventions: Other: quality of life questionnaire

INTERVENTIONS:
Other: quality of life questionnaire — telephone interview to assess mortality and quality of life in the population included in a trial

SUMMARY:
Long term follow up of patients included in a randomized controlled trial evaluating awake prone positioning among patients suffering SARS-CoV2 pneumonia (NCT04358939)

DETAILED DESCRIPTION:
All patients included in the initial trial who survived and were not lost to follow up at 28 days will be invited for a telephone interview to collect data on long term quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients included in the randomized meta-trial evaluating awake prone position versus control among COVID-19 patients on high-flow nasal oxygen therapy (Ehrmann 2021).
* Patients alive at D28
* No opposition to participate in the research which evaluates mortality and quality of life by telephone interview.

Exclusion Criteria:

* Patients lost to follow-up after 28 days.
* Withdrawal of consent from randomized meta-trial by patient
* Vulnerable person: safeguard of justice, curatorship, or guardianship
* Patients refusing to answer telephone questionnaire.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients included in France in the randomized study "High Prone Covid" alive at day 28 (NCT04358939).
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-05-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
EURO QoL 5D 5L quality-of-life score | 2 years after randomization
  Quality of life at last follow-up, beyond 2 years after randomization, assessed by a EURO QoL 5D 5L quality-of-life score

SECONDARY OUTCOMES:
Mortality at last follow-up time beyond 2 years after randomization | an average of 2 years follow up
Assessment of autonomy | an average of 2 years follow up
  Subpart of EURO QoL 5D 5L score
Assessment of mobility | an average of 2 years follow up
  Subpart of EURO QoL 5D 5L score
Assessment of performance of daily activities | an average of 2 years follow up
  Subpart of EURO QoL 5D 5L score
Assessment of pain and discomfort | an average of 2 years follow up
  Subpart of EURO QoL 5D 5L score
Assessment of anxiety and depression | an average of 2 years follow up
  Subpart of EURO QoL 5D 5L score
Number of points on the visual analog scale | an average of 2 years follow up
  Subpart of EURO QoL 5D 5L score
Hospitalisations | an average of 2 years follow up
  Number of new hospitalizations during follow-up period
Family situation | before hospitalization in intensive care unit, then at 12, 24 months and at final follow-up.
  Change of family situation
Employment status | before hospitalization, then at 12, 24 months and at final follow-up.
  Change of employment status
Subgroup analysis: | an average of 2 years follow up
  analysis of primary endpoint, mortality, and subparts of the EURO QoL 5D 5L score in subgroups of patients who were intubated or not during follow-up in the initial meta-assay

CONTACTS AND LOCATIONS:
Locations (1):
- university hospital Tours, Tours, France

IPD SHARING:
Plan to Share IPD: Undecided